CLINICAL TRIAL: NCT02318602
Title: A Multicenter, Open-label, Flexible Dose Study to Assess the Long-term Safety of Pharmaceutical Cannabidiol Oral Solution as an Adjunctive Treatment for Pediatric Subjects With a Treatment-resistant Seizure Disorder Who Complete INS011-14-029 or Part A of INS011-15-054
Brief Title: Cannabidiol Oral Solution as an Adjunctive Treatment for Treatment-resistant Seizure Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INS011-14-030
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Seizures
Keywords: Lennox-Gastaut syndrome; Dravet syndrome; Treatment-resistant seizures
MeSH Terms: conditions — Seizures; Lennox Gastaut Syndrome; Epilepsies, Myoclonic | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Infants (Experimental): Participants 1 to<2 years of age. Participants who completed INS011-14-029 initiated this study on the dose with which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant. The maximum daily dose was 40 mg/kg/day.
  Participants who enrolled from INS011-15-054 continued treatment with the dose at which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  The total daily dose, milligrams per kilograms per day (mg/kg/day), will be evenly split between morning and evening doses (12 hours apart). If tolerability issues arise, the participant's dose may be changed at the investigator's discretion.
  Interventions: Drug: Cannabidiol Oral Solution
- Children (Experimental): Participants 2 to <12 years of age. Participants who completed INS011-14-029 initiated this study on the dose with which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.The maximum daily dose was 40 mg/kg/day.
  Participants who enrolled from INS011-15-054 continued treatment with the dose at which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  The total daily dose (mg/kg/day) will be evenly split between morning and evening doses (12 hours apart). If tolerability issues arise, the participant's dose may be changed at the investigator's discretion.
  Interventions: Drug: Cannabidiol Oral Solution
- Adolescents (Experimental): Participants 12 to <17 years of age. Participants who completed INS011-14-029 initiated this study on the dose with which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant. The maximum daily dose was 40 mg/kg/day.
  Participants who enrolled from INS011-15-054 continued treatment with the dose at which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  The total daily dose (mg/kg/day) will be evenly split between morning and evening doses (12 hours apart). If tolerability issues arise, the participant's dose may be changed at the investigator's discretion.
  Interventions: Drug: Cannabidiol Oral Solution

INTERVENTIONS:
Drug: Cannabidiol Oral Solution — An oral solution containing pharmaceutical grade cannabidiol (nonplant-based).

SUMMARY:
This is a multicenter, open-label trial to assess the long-term safety and efficacy of Cannabidiol Oral Solution as adjunctive therapy for pediatric participants with treatment-resistant seizure disorders, including Lennox-Gastaut syndrome (LGS) or Dravet syndrome (DS). All participants have rolled over from previous trials: INS011-14-029 (NCT02324673) and INS011-15-054 (NCT02551731).

ELIGIBILITY:
Inclusion Criteria:

* Completed activities through Day 11 in INS011-14-029 or Part A (Visit 6) INS011-15-054
* Informed consent/assent (as applicable) was voluntarily provided by the participant and/or parent(s)/caregiver(s) in accordance with applicable laws, regulations, and local requirements
* Is medically stable with no anticipated changes in chronic medications in the opinion of the Investigator
* Continues to meet protocol-specified criteria for qualification and contraception, including treatment-resistant seizure disorder
* In the opinion of the Investigator, the subject and/or parent(s)/caregiver(s) are able to continue keeping accurate seizure diaries

Exclusion Criteria:

* Inadequate supervision by parent(s)/caregiver(s)
* History or current use of dietary supplements, drugs or over-the counter medications outside protocol-specified parameters
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
  3. the analysis of results

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neha Parikh, Study Director — INSYS Therapeutics Inc
Locations (11):
- United States (11):
  - University of California San Francisco Medical Center, San Francisco, California
  - Miami Children's Hospital, Miami, Florida
  - Child Neurology Center - NW F, Pensacola, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Clinical Research Center of Nevada LLC, Las Vegas, Nevada
  - Oregon Health Services University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Texas Scottish Rite Hospital for Children, Dallas, Texas
  - Granger Medical Clinic, Riverton, Utah
  - Mary Bridge Children's Hospital, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Infants: Participants 1 to <2 years of age. Participants who completed INS011-14-029 initiated this study on the dose with which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  Participants who enrolled from INS011-15-054 continued treatment with the dose at which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  The total daily dose (mg/kg/day) will be evenly split between morning and evening doses (12 hours apart). If tolerability issues arise, the participant's dose may be changed at the investigator's discretion.
- Children: Participants 2 to <12 years of age. Participants who completed INS011-14-029 initiated this study on the dose with which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  Participants who enrolled from INS011-15-054 continued treatment with the dose at which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  The total daily dose (mg/kg/day) will be evenly split between morning and evening doses (12 hours apart). If tolerability issues arise, the participant's dose may be changed at the investigator's discretion.
- Adolescents: Participants 12 to ≤17 years of age. Participants who completed INS011-14-029 initiated this study on the dose with which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  Participants who enrolled from INS011-15-054 continued treatment with the dose at which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  The total daily dose (mg/kg/day) will be evenly split between morning and evening doses (12 hours apart). If tolerability issues arise, the participant's dose may be changed at the investigator's discretion.
Period: Overall Study
Arm/Group | Infants | Children | Adolescents
Started | 9 | 26 | 17
Completed | 8 | 22 | 15
Not Completed | 1 | 4 | 2
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Guardian decision to withdraw | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Infants: Participants 1 to <2 years of age.Participants who completed INS011-14-029 initiated this study on the dose with which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  Participants who enrolled from INS011-15-054 continued treatment with the dose at which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  The total daily dose (mg/kg/day) will be evenly split between morning and evening doses (12 hours apart). If tolerability issues arise, the participant's dose may be changed at the investigator's discretion.
- Children: Participants 2 to <12 years of age.Participants who completed INS011-14-029 initiated this study on the dose with which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  Participants who enrolled from INS011-15-054 continued treatment with the dose at which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  The total daily dose (mg/kg/day) will be evenly split between morning and evening doses (12 hours apart). If tolerability issues arise, the participant's dose may be changed at the investigator's discretion.
- Adolescents: Participants 12 to <17 years of age.Participants who completed INS011-14-029 initiated this study on the dose with which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  Participants who enrolled from INS011-15-054 continued treatment with the dose at which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  The total daily dose (mg/kg/day) will be evenly split between morning and evening doses (12 hours apart). If tolerability issues arise, the participant's dose may be changed at the investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Infants | Children | Adolescents | Total
Number analyzed (Participants) | 9 | 26 | 17 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1.00 (0.00) | 6.7 (2.84) | 13.9 (1.58) | 8.1 (5.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 9 | 24
  Male | 5 | 15 | 8 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 7 | 24 | 16 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 2 | 0 | 2
  White | 8 | 19 | 16 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 26 | 17 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An Adverse Event (AE) is any untoward medical occurrence in a subject administered a pharmaceutical product. It does not necessarily have a causal relationship with this treatment.
Time Frame: Up to Week 50
Measure: Number; unit: Percentage of participants
Groups:
- All Participants: All participants who participated in the study.
Arm/Group | Infants | Children | Adolescents | All Participants
Number analyzed (Participants) | 9 | 26 | 17 | 52
Percentage of participants | 88.9 | 92.3 | 88.2 | 90.4

2. Primary Outcome: Percentage of Participants With Serious Adverse Events
Description: A serious adverse event is any untoward medical occurrence ( whether considered to be related to investigational product or not) that at any dose results in death, is life threatening, requires inpatient hospitalization, results in disability/incapacity, is a congenital abnormality/ birth defect, or medically significant as determined by an investigator.
Time Frame: Up to Week 50
Measure: Number; unit: Percentage of participants
Arm/Group | Infants | Children | Adolescents | All Participants
Number analyzed (Participants) | 9 | 26 | 17 | 52
Percentage of participants | 77.8 | 38.5 | 0 | 32.7

3. Primary Outcome: Percentage of Participants With Clinically Significant Change From Baseline in Laboratory Values
Description: Laboratory values include chemistry and hematology, and urinary analysis.
Time Frame: Up to Week 50
Measure: Number; unit: Percentage of participants
Arm/Group | Infants | Children | Adolescents
Number analyzed (Participants) | 9 | 26 | 17
Percentage of participants
  Hematology | 0 | 0 | 0
  Blood Chemistry | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Findings
Time Frame: Up to Week 48
Measure: Number; unit: Percentage of participants
Groups:
- Infants: Participants 1 to<2 years of age. Participants who completed INS011-14-029 initiated this study on the dose with which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  Participants who enrolled from INS011-15-054 continued treatment with the dose at which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  The total daily dose (mg/kg/day) will be evenly split between morning and evening doses (12 hours apart). If tolerability issues arise, the participant's dose may be changed at the investigator's discretion.
- Adolescents: Participants 12 to <17 years of age. Participants who completed INS011-14-029 initiated this study on the dose with which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  Participants who enrolled from INS011-15-054 continued treatment with the dose at which they were being treated previously, and dose modifications were made at the Investigator's discretion if tolerability or efficacy issues were observed for a particular participant.
  The total daily dose (mg/kg/day) will be evenly split between morning and evening doses (12 hours apart). If tolerability issues arise, the participant's dose may be changed at the investigator's discretion.
Arm/Group | Infants | Children | Adolescents
Number analyzed (Participants) | 9 | 26 | 17
Percentage of participants | 0 | 0 | 0

5. Primary Outcome: Percentage of Participants With Clinically Significant Change From Baseline in Vital Signs
Time Frame: Up to Week 50
Measure: Number; unit: Percentage of participants
Arm/Group | Infants | Children | Adolescents
Number analyzed (Participants) | 9 | 26 | 17
Percentage of participants | 0 | 0 | 0

6. Primary Outcome: Change From Baseline in Trough Plasma Levels of Cannabidiol and Its 7-OH Metabolite
Time Frame: Up to Week 50
Population: Insufficient data was collected to perform study analysis.
Arm/Group | Infants | Children | Adolescents
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Vineland Adaptive Behavior Scales (VABS)
Description: The Vineland Adaptive Behavior Scales measures the personal and social skills of individuals from birth through adulthood. Because adaptive behavior refers to an individual's typical performance of the day-to-day activities required for personal and social sufficiency, these scales assess what a person actually does, rather than what he or she is able to do.
  The Vineland Adaptive Behavior Scales, Second Edition (Survey Interview Form) is a measure of adaptive behavior in children, adolescents and adults. It yields an overall standard score (Adaptive Behavior Composite, ABC) and age standard scores in four domains. The 4 domains are Communication, Daily Living Skills, Motor Skills, and Maladaptive Behaviour Index. ABC scores have a mean of 100 and a standard deviation of 15 (range = 20 to 160). Higher scores suggest a higher level of adaptive functioning. A rise in standard scores from Baseline indicates improvement.
  The VABS will be completed for all participants.
Time Frame: Up to Week 48
Population: The Safety Analysis Population (SAF) consisted of all participants in the enrolled population group (ENR) who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infants | Children | Adolescents
Number analyzed (Participants) | 9 | 26 | 17
Score on a scale
  Communication: Expressive (Day 1) | 6.8 (7.34) | 40.4 (37.53) | 40.3 (42.76)
  Communication: Expressive (Week 36): number analyzed (Participants) | 7 | 17 | 12
  Communication: Expressive (Week 36) | 8.3 (9.03) | 51.7 (41.79) | 36.0 (41.63)
  Communication: Expressive (Week 48): number analyzed (Participants) | 8 | 25 | 13
  Communication: Expressive (Week 48) | 9.9 (9.30) | 48.6 (38.91) | 34.3 (40.62)
  Communication: Receptive (Day 1) | 6.0 (7.35) | 17.4 (13.10) | 18.8 (14.88)
  Communication: Receptive (Week 36): number analyzed (Participants) | 7 | 17 | 12
  Communication: Receptive (Week 36) | 8.6 (7.23) | 21.1 (13.15) | 15.7 (15.95)
  Communication: Receptive (Week 48): number analyzed (Participants) | 8 | 25 | 13
  Communication: Receptive (Week 48) | 11.5 (8.73) | 20.6 (13.15) | 16.8 (14.62)
  Communication: Written (Day 1): number analyzed (Participants) | 4 | 24 | 17
  Communication: Written (Day 1) | 0.0 (0.00) | 9.2 (13.47) | 12.9 (17.09)
  Communication: Written (Week 36): number analyzed (Participants) | 3 | 16 | 12
  Communication: Written (Week 36) | 1.3 (2.31) | 11.8 (15.98) | 12.8 (17.33)
  Communication: Written (Week 48): number analyzed (Participants) | 7 | 25 | 13
  Communication: Written (Week 48) | 0.0 (0.00) | 10.8 (13.88) | 10.5 (17.15)
  Daily Living Skills: Community (Day 1): number analyzed (Participants) | 9 | 26 | 16
  Daily Living Skills: Community (Day 1) | 0.4 (1.33) | 13.8 (18.62) | 19.1 (26.03)
  Daily Living Skills: Community (Week 36): number analyzed (Participants) | 7 | 17 | 12
  Daily Living Skills: Community (Week 36) | 0.6 (1.51) | 17.8 (19.99) | 18.8 (26.58)
  Daily Living Skills: Community (Week 48): number analyzed (Participants) | 8 | 25 | 13
  Daily Living Skills: Community (Week 48) | 1.0 (2.14) | 16.6 (21.29) | 18.8 (29.07)
  Daily Living Skills: Domestic (Day 1) | 0.4 (1.33) | 9.1 (11.85) | 9.7 (15.70)
  Daily Living Skills: Domestic (Week 36): number analyzed (Participants) | 7 | 17 | 12
  Daily Living Skills: Domestic (Week 36) | 0.9 (2.27) | 9.6 (12.45) | 10.7 (16.42)
  Daily Living Skills: Domestic (Week 48): number analyzed (Participants) | 8 | 24 | 13
  Daily Living Skills: Domestic (Week 48) | 0.8 (2.12) | 9.9 (13.43) | 9.2 (15.71)
  Daily Living Skills: Personal (Day 1): number analyzed (Participants) | 9 | 26 | 16
  Daily Living Skills: Personal (Day 1) | 3.6 (6.65) | 31.7 (29.37) | 28.6 (27.98)
  Daily Living Skills: Personal (Week 36): number analyzed (Participants) | 7 | 17 | 12
  Daily Living Skills: Personal (Week 36) | 5.0 (8.93) | 39.2 (29.64) | 26.2 (29.19)
  Daily Living Skills: Personal (Week 48): number analyzed (Participants) | 8 | 25 | 13
  Daily Living Skills: Personal (Week 48) | 5.6 (8.09) | 36.2 (30.66) | 25.4 (29.78)
  Socialization: Coping Skills (Day 1): number analyzed (Participants) | 9 | 26 | 16
  Socialization: Coping Skills (Day 1) | 2.1 (2.67) | 14.6 (18.34) | 16.9 (20.33)
  Socialization: Coping Skills (Week 36): number analyzed (Participants) | 7 | 17 | 12
  Socialization: Coping Skills (Week 36) | 2.6 (3.99) | 16.2 (16.37) | 16.7 (20.81)
  Socialization: Coping Skills (Week 48): number analyzed (Participants) | 8 | 25 | 13
  Socialization: Coping Skills (Week 48) | 3.1 (4.32) | 15.0 (17.08) | 15.9 (20.63)
  Socialization: Interpersonal Relationships (Day 1) | 9.4 (10.14) | 28.9 (22.93) | 31.1 (25.41)
  Socialization: Interpersonal Relationships (Wk 36): number analyzed (Participants) | 7 | 17 | 12
  Socialization: Interpersonal Relationships (Wk 36) | 11.9 (10.67) | 35.7 (21.85) | 25.8 (22.75)
  Socialization: Interpersonal Relationships (Wk 48): number analyzed (Participants) | 8 | 25 | 13
  Socialization: Interpersonal Relationships (Wk 48) | 14.0 (12.62) | 33.3 (22.67) | 26.7 (24.35)
  Socialization: Play and Leisure Time (Day 1): number analyzed (Participants) | 9 | 26 | 16
  Socialization: Play and Leisure Time (Day 1) | 5.3 (9.53) | 20.5 (20.11) | 19.7 (20.62)
  Socialization: Play and Leisure Time (Week 36): number analyzed (Participants) | 7 | 17 | 12
  Socialization: Play and Leisure Time (Week 36) | 6.6 (10.55) | 24.4 (19.77) | 19.6 (22.71)
  Socialization: Play and Leisure Time (Week 48): number analyzed (Participants) | 8 | 24 | 13
  Socialization: Play and Leisure Time (Week 48) | 6.4 (10.16) | 21.8 (18.96) | 17.9 (22.66)
  Motor Skills: Fine (Day 1) | 4.2 (9.72) | 26.7 (27.29) | 23.1 (26.20)
  Motor Skills: Fine (Week 36): number analyzed (Participants) | 7 | 17 | 11
  Motor Skills: Fine (Week 36) | 5.1 (12.29) | 33.6 (27.38) | 20.9 (24.32)
  Motor Skills: Fine (Week 48): number analyzed (Participants) | 8 | 25 | 13
  Motor Skills: Fine (Week 48) | 6.0 (8.67) | 32.2 (27.56) | 24.0 (25.21)
  Motor Skills: Gross (Day 1) | 8.0 (18.45) | 42.5 (31.90) | 31.0 (29.57)
  Motor Skills: Gross (Week 36): number analyzed (Participants) | 7 | 17 | 11
  Motor Skills: Gross (Week 36) | 11.0 (22.96) | 46.5 (32.43) | 31.9 (26.74)
  Motor Skills: Gross (Week 48): number analyzed (Participants) | 8 | 25 | 13
  Motor Skills: Gross (Week 48) | 12.8 (22.42) | 46.6 (32.44) | 33.3 (29.03)
  Maladaptive Behavior Index: Externalizing (Day 1): number analyzed (Participants) | 0 | 26 | 17
  Maladaptive Behavior Index: Externalizing (Day 1) |  | 3.5 (3.51) | 3.5 (3.10)
  Maladaptive Behavior Index: Externalizing (Wk 36): number analyzed (Participants) | 2 | 17 | 12
  Maladaptive Behavior Index: Externalizing (Wk 36) | 0.0 (0.00) | 4.5 (4.81) | 3.1 (3.42)
  Maladaptive Behavior Index: Externalizing (Wk 48): number analyzed (Participants) | 4 | 25 | 13
  Maladaptive Behavior Index: Externalizing (Wk 48) | 0.0 (0.00) | 4.4 (4.10) | 2.2 (2.95)
  Maladaptive Behavior Index: Internalizing (Day 1): number analyzed (Participants) | 0 | 26 | 16
  Maladaptive Behavior Index: Internalizing (Day 1) |  | 5.2 (4.01) | 3.6 (3.24)
  Maladaptive Behavior Index: Internalizing (Wk 36): number analyzed (Participants) | 2 | 17 | 12
  Maladaptive Behavior Index: Internalizing (Wk 36) | 0.0 (0.00) | 5.4 (3.06) | 3.7 (3.63)
  Maladaptive Behavior Index: Internalizing (Wk 48): number analyzed (Participants) | 4 | 25 | 13
  Maladaptive Behavior Index: Internalizing (Wk 48) | 1.0 (2.00) | 5.3 (4.10) | 3.6 (3.62)
  Maladaptive Behavior Index: MBI Score (Day 1): number analyzed (Participants) | 0 | 26 | 16
  Maladaptive Behavior Index: MBI Score (Day 1) |  | 14.8 (7.53) | 13.0 (8.75)
  Maladaptive Behavior Index: MBI Score (Week 36): number analyzed (Participants) | 2 | 17 | 12
  Maladaptive Behavior Index: MBI Score (Week 36) | 0.0 (0.00) | 16.6 (8.65) | 10.8 (9.04)
  Maladaptive Behavior Index: MBI Score (Week 48): number analyzed (Participants) | 4 | 24 | 13
  Maladaptive Behavior Index: MBI Score (Week 48) | 1.0 (2.00) | 16.1 (9.17) | 10.2 (8.47)
  Maladaptive Behavior Index: Other (Day 1): number analyzed (Participants) | 0 | 26 | 17
  Maladaptive Behavior Index: Other (Day 1) |  | 6.2 (4.17) | 6.2 (4.76)
  Maladaptive Behavior Index: Other (Week 36): number analyzed (Participants) | 2 | 17 | 12
  Maladaptive Behavior Index: Other (Week 36) | 0.0 (0.00) | 6.7 (4.01) | 4.1 (3.60)
  Maladaptive Behavior Index: Other (Week 48): number analyzed (Participants) | 4 | 24 | 13
  Maladaptive Behavior Index: Other (Week 48) | 0.0 (0.00) | 6.5 (3.30) | 4.3 (3.88)

8. Secondary Outcome: Number of Participants With a Positive Response on the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: For subjects 7 years of developmental age or older, the Columbia-Suicide Severity Rating Scale (C-SSRS) will be administered to access suicidality. The appropriate adult version will be used in subjects 12 years of (developmental) age and older. The investigator will determine the participant's developmental age.
Time Frame: Up to Week 50
Measure: Count of Participants; unit: Participants
Arm/Group | Infants | Children | Adolescents
Number analyzed (Participants) | 9 | 26 | 17
Participants
  Suicidal Ideation | 0 | 0 | 0
  Suicidal Behavior | 0 | 0 | 0

9. Other Pre Specified Outcome: Clinical Global Impression of Severity (CGI-S)
Description: The severity of the participant's illness is rated on a seven-point scale, where 1=normal, not at all ill, and 7=among the most extremely ill patients. This rating is based upon observed and reported symptoms, behavior, and function in the past seven days. The score reflects the average severity level across the seven days.
  The CGI-S will be completed for all participants, regardless of chronological and developmental age.
Time Frame: through study completion, up to 48 weeks or marketing approval, whichever is earlier
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Impact of Pediatric Epilepsy Scale (IPES)
Description: The IPES assesses the impact on academic achievement, participation in activities, health, relationships with family and with peers and siblings, social activities, self-esteem, and the caregiver's hopes for their child's future. It takes about 3 minutes for the parent to complete. Each of the 11 items is given a severity score of 0 (not at all) to 3 (a lot). The higher the score, the higher is the impact of epilepsy on that item. The highest total score possible is 33 (range 0-33).
  The Impact of Pediatric Epilepsy Scale (IPES) is validated for subjects who are 2 to 16 years of age. Due to developmental delay characteristic of the study population, subjects through 18 years of chronological age will complete the IPES. Subjects over 18 years of chronological age will not complete the IPES.
Time Frame: through study completion, up to 48 weeks or marketing approval, whichever is earlier
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Clinical Global Impression of Improvement (CGI-I)
Description: The participant's overall clinical condition is compared to the one week period just before the start of medication (the baseline visit). The participant's condition is compared to the patient's condition at admission to the project [prior to starting treatment] on a 7-point scale, where 1=very much improved since the initiation of treatment; and 7=very much worse since the initiation of treatment.
  The CGI-I will be completed for all participants, regardless of chronological and developmental age.
Time Frame: through study completion, up to 48 weeks or marketing approval, whichever is earlier
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change From Baseline in Frequency of Seizures as a Measure of Seizure Control
Time Frame: through study completion, up to 48 weeks or marketing approval, whichever is earlier
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to Week 50
Arm/Group | Infants | Children | Adolescents
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/26 | 0/17
Serious Adverse Events (participants affected / at risk) | 7/9 | 10/26 | 0/17
Other Adverse Events (participants affected / at risk) | 8/9 | 24/26 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infants (N=9) | Children (N=26) | Adolescents (N=17)
Seizure (Nervous system disorders) | 5 | 5 | 0
Status epilepticus (Nervous system disorders) | 2 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Change in seizure presentation (Nervous system disorders) | 1 | 0 | 0
Adenovirus infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Physical assault (Social circumstances) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infants (N=9) | Children (N=26) | Adolescents (N=17)
Upper respiratory tract infection (Infections and infestations) | 1 | 6 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3 | 1
Otitis media (Infections and infestations) | 0 | 5 | 0
Influenza (Infections and infestations) | 1 | 3 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0
Mycoplasma infection (Infections and infestations) | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Vestibulitis (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Seizure (Nervous system disorders) | 4 | 9 | 3
Somnolence (Nervous system disorders) | 2 | 4 | 1
Ataxia (Nervous system disorders) | 0 | 2 | 0
Epilepsy (Nervous system disorders) | 1 | 1 | 0
Status epilepticus (Nervous system disorders) | 2 | 0 | 0
Change in seizure presentation (Nervous system disorders) | 1 | 0 | 0
Clumsiness (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Fontanelle bulging (Nervous system disorders) | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1
Postictal paralysis (Nervous system disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 5 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 1
Irritability (Psychiatric disorders) | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Flat affect (Psychiatric disorders) | 0 | 0 | 1
Head banging (Psychiatric disorders) | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 2
Constipation (Gastrointestinal disorders) | 0 | 4 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 3 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 4 | 0
Device expulsion (General disorders) | 1 | 0 | 0
Device failure (General disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Weight increased (Investigations) | 0 | 4 | 0
Human rhinovirus test positive (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 6 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Pulmonary valve incompetence (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT02318602/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT02318602/SAP_001.pdf